CLINICAL TRIAL: NCT01917188
Title: Promoting Patient-Centered Care Through a Heart Failure Simulation Study
Acronym: HF SIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: Intermountain Research and Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1024572
Record Dates: First submitted 2013-08-01; First posted 2013-08-06 (Estimated); Results first posted 2019-01-16 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2018-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Full simulation and education (Active Comparator): Patients who will receive full simulation and education session prior to discharge.
  Interventions: Behavioral: Full simulation and education
- See simulation room, usual education (Other): Patients will be shown the simulation room prior to discharge but will only receive usual education.
  Interventions: Behavioral: See simulation room, usual education
- Usual care (No Intervention): Patients will receive usual care by bedside nurse.

INTERVENTIONS:
Behavioral: Full simulation and education
  Arms: Full simulation and education
Behavioral: See simulation room, usual education
  Arms: See simulation room, usual education

SUMMARY:
The initial aim of this study will be to assess current methods of heart failure (HF) patient education in terms of patient satisfaction, level of preparedness for home, and care provider satisfaction. The second aim will be to design and create a "living with HF at home" simulation session. The third aim will test the hypothesis that hospitalized HF patients who receive education in a simulation room in addition to usual HF education will have improved qualitative and quantitative outcomes as compared to those who do not receive the additional education support.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 years of age.
2. Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.
3. Documentation of HF of any etiology based on clinical assessment of the Primary Investigator, using standard-of-care criteria for diagnosis.
4. Heart failure of either preserved or reduced ventricular function.

Exclusion Criteria:

1. Patients requiring ICU monitoring
2. LVAD candidate/recipient
3. Cardiac transplant candidate/recipient
4. Confusion
5. Sepsis
6. Terminal illness (other than HF) with expected survival of less than 1 year
7. Enrollment or planned enrollment in another randomized clinical trial during this hospitalization
8. Inability to comply with planned study procedures
9. Active illicit drug use
10. Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study.
11. Other conditions that in the opinion of the Primary Investigator may increase risk to the subject and/or compromise the quality of the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-11; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kismet D Rasmusson, FNP-BC, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Full Simulation and Education: Patients who will receive full simulation and education session prior to discharge.
  Full simulation and education
- See Simulation Room, Usual Education: Patients will be shown the simulation room prior to discharge but will only receive usual education.
  See simulation room, usual education
Period: Overall Study
Arm/Group | Full Simulation and Education | See Simulation Room, Usual Education | Usual Care
Started | 29 | 23 | 20
Completed | 17 | 17 | 11
Not Completed | 12 | 6 | 9

BASELINE CHARACTERISTICS:
Population: Only included those who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Full Simulation and Education | See Simulation Room, Usual Education | Usual Care | Total
Number analyzed (Participants) | 17 | 17 | 11 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (13) | 67.9 (8.2) | 62.7 (11.6) | 65.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 2 | 1 | 11
  Male | 9 | 15 | 10 | 34

OUTCOME MEASURES:

1. Primary Outcome: Mean Differences in Minnesota Living With Heart Failure Questionnaire (MLHFQ) Results
Description: The mean differences in heart failure knowledge (from study enrollment to the 30 day study follow up) in each of the arms as assessed by the MLHFQ. Lower scores indicate improvement and a better health-related quality of life (HRQoL).
  The MLHFQ is a self-administered questionnaire for patients with HF, comprising 21 items rated on six-point Likert scales, representing different degrees of impact of HF on HRQoL, from 0 (none) to 5 (very much). It provides a total score (range 0-105, from best to worst HRQoL), as well as scores for two dimensions, physical (8 items, range 0-40) and emotional (5 items, range 0-25). The other eight items (of the total of 21) are only considered for the calculation of the total score.
Time Frame: 30 days
Population: Only a small number of people completed and returned the quiz.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Full Simulation and Education | See Simulation Room, Usual Education | Usual Care
Number analyzed (Participants) | 16 | 17 | 11
score on a scale
  Total Score Difference | -4.69 (35.06) | -26.59 (28.25) | -29.36 (35.69)
  Physical Score Difference | -4.31 (15.25) | -13.24 (11.51) | -15.09 (14.58)
  Emotional Score Difference | -0.88 (8.60) | -6.59 (8.28) | -5.27 (8.88)

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Full Simulation and Education | See Simulation Room, Usual Education | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/29 | 1/23 | 1/20
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/23 | 1/20
Other Adverse Events (participants affected / at risk) | 1/29 | 0/23 | 1/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Simulation and Education (N=29) | See Simulation Room, Usual Education (N=23) | Usual Care (N=20)
Knee wound dehiscence (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Acute traumatic left knee wound dehiscence.
Subarachnoid hemorrhage after a fall (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Full Simulation and Education (N=29) | See Simulation Room, Usual Education (N=23) | Usual Care (N=20)
lightheaded (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes